CLINICAL TRIAL: NCT04769349
Title: Effectiveness of Supportive Housing on COVID-19 Related Outcomes for People Experiencing Homelessness
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Benjamin F. Henwood, Associate Professor, University of Southern California
Other Study IDs: UP-20-01081
Record Dates: First submitted 2021-02-09; First posted 2021-02-24 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Housing; Covid19; Mental Health; Physical Health; Social Interaction; Healthcare
MeSH Terms: conditions — COVID-19; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to understand the comparative effectiveness of two PSH models (PB-PSH and SS-PSH) on quality of life and COVID-19 related health behaviors by following for 6 months a cohort of 800 PEH who have been placed in either PB (n=400) or SS (n=400). In a natural observational experiment, participants will complete 6 monthly mobile-based questionnaires exploring quality of life including physical, mental, social, and housing/environmental health, COVID-19 prevention practices (i.e., handwashing, social distancing, face covering), and past-30-day healthcare utilization. A sub-sample of 40 participants living in both PB-PSH and SS-PSH will be qualitatively interviewed longitudinally to help contextualize quantitative findings. Focus groups will also be conducted with providers of PSH and qualitative interviews will be conducted with other key stakeholders to understand perspectives on the challenges of implementing and sustaining COVID-19 related prevention practices while maintaining a continuity of care.

DETAILED DESCRIPTION:
This study will aim to understand the comparative effectiveness of PB-PSH and SS-PSH on patient-centered quality of life, health care utilization, and health behaviors that will reduce COVID-19 risk by following a diverse sample of 800 PEH who are placed in PB-PSH (n = 400) or SS-PSH (n = 400) for 6 months. Barriers and facilitators will also be identified that may affect PSH implementation during the pandemic and its aftermath. The specific aims are:

Aim 1: To test the comparative effectiveness of PB-PSH and SS-PSH on COVID-19-related health behaviors (COVID-19-related personal health practices including social distancing) for PEH over time.

Aim 2: To test the comparative effectiveness of PB-PSH and SS-PSH on patient-centered quality of life (i.e., general life satisfaction; physical, mental, social, and environmental health) for PEH over time.

Aim 3: To test the comparative effectiveness of PB-PSH and SS-PSH on health care utilization health behaviors and unmet need for care for physical health, mental health, substance use disorders, for PEH over time.

Aim 4: To contextualize quantitative findings through longitudinal qualitative inquiry with 40 participants, purposively sampled from PB-PSH and SS-PSH, based on whether they are following social distancing guidelines.

Aim 5: To understand service providers, policy makers, and other stakeholders perspectives on challenges of implementing and sustaining COVID-19-related prevention practices and continuity of care in PSH.

ELIGIBILITY:
Inclusion Criteria:

* adults (aged 18+) with recent (past 12 months) lived experience with homelessness
* approved for PSH
* proficient in English
* able to provide informed consent

Exclusion Criteria:

* aged younger than 18
* not approved for PSH
* not proficient in English
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 800 adults experiencing homelessness who have been approved for permanent supportive housing (PSH) in Los Angeles
Sampling Method: Non-Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Life Satisfaction | Change of Life satisfaction from baseline to 6 months
  The NIH Toolbox item Bank v2.0 contains 10 items and will be utilized for participants to self-rate their life satisfaction
Quality of physical health | Change in quality of physical health from baseline to 6 months
  Self-rated physical health and frequency/quantity of health-related activities will be assessed with the PROMIS Global Health Scale Version 1.2. Scores range from 1-10, with higher scores reflecting better functioning.
Degree of mental health symptomatology | Change in symptomatology from baseline to 6 months
  The PROMIS will also be utilized to assess self-rated frequency the participant is bothered by mental health symptoms. The lowest possible score is 8 and the highest possible score is 40. Higher scores reflect more problematic symptomatology.
Social Isolation | Change in social isolation from baseline to 6 months
  The PROMIS will be utilized to assess social isolation including perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others. Scores range from 6 to 40 with higher scores representing increased perceptions of isolation.
Housing Environment | Change in satisfaction with housing environment from baseline to 6 months
  The Housing Environment Scale will assess residential satisfaction and neighborhood quality/safety. There are 5 subscales assessing the following: physical quality of the home, perceived quality of the neighborhood, perceived social climate in neighborhood, physical quality of home, and the physical quality of the neighborhood. Scales contain a range of 14 to 17 items with scores that range from 14 to 85 with higher scores representing increased satisfaction with environment.

SECONDARY OUTCOMES:
COVID-19 Prevention practices | Change in use of prevention practices from baseline to 6 months
  The NIH Disaster Research Response Platform will assess participant frequency of handwashing, social distancing, and use of face covering.
Healthcare Utilization | Change in utilization from baseline to 6 months
  Participants will record their past 30-day use of physical and mental health treatment, social services, and support provided by the permanent supportive housing program

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Henwood, Principal Investigator — University of Southern California
Locations (1):
- Los Angeles Homeless Services Authority (LAHSA), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henwood BF, Kuhn R, Padwa H, Ijadi-Maghsoodi R, Corletto G, Lawton A, Chien J, Bluthenthal R, Cousineau MR, Chinchilla M, Tran Smith B, Vickery KD, Harris T, Patanwala M, Akabike W, Gelberg L. Investigating the Comparative Effectiveness of Place-Based and Scatter-Site Permanent Supportive Housing for People Experiencing Homelessness During the COVID-19 Pandemic: Protocols for a Mixed Methods, Prospective Longitudinal Study. JMIR Res Protoc. 2023 Apr 28;12:e46782. doi: 10.2196/46782. PMID 37115590